CLINICAL TRIAL: NCT05600400
Title: Improving Sexual Quality of Life - A Phase 2 Randomized Controlled Trial of Two Versus Five Stereotactic MRI-Guided Ablative Radiotherapy Treatments for Prostate Cancer
Brief Title: Improving Sexual Quality of Life - Randomized Trial of Two vs Five MRI Guided SABR Treatments for Prostate Cancer
Acronym: iSMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Prostate Cure Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. Danny Vesprini, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iSMART
Record Dates: First submitted 2022-10-12; First posted 2022-10-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Cancer of Prostate; Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 fraction SBRT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Two weekly fractions of 13.5 Gy
  Interventions: Radiation: Stereotactic Ablative Body Radiation
- Arm 2 (Active Comparator): Five every other day fractions of 8 Gy
  Interventions: Radiation: Stereotactic Ablative Body Radiation

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiation — 2 Fraction
  Other Names: SBRT

SUMMARY:
Prostate Stereotactic ablative body radiotherapy (SABR) is an established technique that delivers radiation in a non-invasive approach for men with prostate cancer. The treatment regimen is given in total of 5 fractions with one treatment per day at every other day or weekly sessions. Ultra-hypofractionated radiotherapy (UHRT) is an emerging monotherapy for localized prostate cancer however, several trials have observed demonstrating superior biochemical control of a two-fraction (HDR) over single-fraction approach. The study aims to compare an experimental shorter course of prostate ultra-hypofractionated radiotherapy (UHRT) that will deliver what is expected to be an equivalent amount of radiation as given in the standard 5 treatment regimen. UHRT is given in 2 treatments with one treatment a week for 2 consecutive weeks.

DETAILED DESCRIPTION:
Ultra-hypofractionated radiotherapy (UHRT) is an emerging monotherapy for localized prostate cancer. From a radiobiological standpoint, fewer fractions and higher doses per fraction takes greater advantage of the low α/β ratio of prostate cancer to improve the therapeutic ratio, most recently estimated at 1.6 based on 14 randomized controlled trials.Highly conformal delivery of large doses per fraction can be achieved with either high dose rate (HDR) brachytherapy or with stereotactic ablative radiotherapy (SABR).

Several trials have explored HDR as monotherapy, from 6-fractions to a single-fraction approach. Sunnybrook recently published a randomized trial of HDR monotherapy demonstrating superior biochemical control of a two-fraction over single-fraction approach. These and other data have informed the design of a phase III randomized controlled trial comparing two-fraction HDR monotherapy to low dose rate (LDR) brachytherapy in patients with intermediate risk prostate cancer (NCT02960087) coordinated by the Canadian Clinical Trails Group (PR19). The investigators have shown that 2 fraction SABR has equivalent efficacy and tolerability to 2 fraction HDR but SABR does not require general anesthesia, is less invasive and cheaper.

UHRT is also supported by phase III data, including a large non-inferiority randomized trial (HYPO-RT-PC) demonstrating similar biochemical control with a 7-fraction versus conventionally-fractionated regimen. The non-inferiority PACE-B trial comparing 5-fraction SABR to conventionally-fractionated or moderately hypofractionated RT has demonstrated similar acute toxicity with use of contemporary SABR planning techniques. Sunnybrook has also conducted several iterative clinical trials testing increasingly hypofractionated external beam radiotherapy. The investigators observed in parallel cohort studies that 5 fractions of UHRT and 2 fractions of UHRT with a patented immobilization device (GU-Lok) had equal effectiveness but better tolerability with the 2 fraction technique. As this was a post hoc analysis, this study aims to validate those findings.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate adenocarcinoma (centrally reviewed)
2. Low or favorable intermediate risk disease. Patient must meet one of the following categories:

   * Low risk - T1-T2b, grade group 1, AND PSA < 10 ng/ml;
   * Favorable risk

     1. Only one of the following intermediate risk factors - cT2c, grade group 2, or PSA 10-20 ng/ml; or
     2. Grade group 3 AND PSA < 20, AND <cT2c AND absolute percentage pattern 4/5 is <10%

Exclusion Criteria:

1. Androgen deprivation therapy (LHRH-agonists or antiandrogens) given or planned
2. Prior pelvic radiotherapy
3. Anticoagulation medication (if unsafe to discontinue for gold seed insertion)
4. Diagnosis of bleeding diathesis
5. Large prostate (>90cm3) on imaging
6. Immunosuppressive medications
7. Inflammatory bowel disease
8. Presence of dual hip prostheses
9. Contraindications to having MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Prostate Cancer Patient's Quality of Life Function will be measured to determine change in Quality of life function from baseline to 5 years beyond treatment. | Change in patient Quaity of Life will be asseses from Before treatment (Baseline); week 1, 4 and 13; month 6 and every 6 months for 5 years
  Expanded Prostate Cancer Index Composite questionnaires will be scored and analyzed to determine change in Quality of life function from baseline

SECONDARY OUTCOMES:
Toxicity in patients | Before treatment (Baseline); week 1, 4 and 13; month 6 and every 6 months for 5 years
  Incidence of acute Gastrointestinal (GI) and Genitourinary (GU) complications using CTCAE v4
Proportion of patients with 4 year PSA value of <0.4 ng/ml | Before treatment (Baseline); months 3 and 6; and every 6 months for 5 years
  Proportion of patients with 4 year PSA value of <0.4 ng/ml
Biochemical Control in Prostate Patients | Before treatment (Baseline); months 3 and 6; and every 6 months for 5 years
  5 year biochemical failure rates using Phoenix definition (as nadir PSA +2ng/mL)
Salvage Therapy Rate | 5 years
  Analysis of prostate patients requiring salvage treatment using Androgen Deprivation Therapy, surgery or brachytherapy
Health Utilities Outcome | 5 years
  Analysis of patient reported outcome using EQ-5D-5L
Health Utilities Outcome | 5 years
  Analysis of patient reported outcome using PORPUS-U

CONTACTS AND LOCATIONS:
Overall Officials: Danny Vesprini, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No